CLINICAL TRIAL: NCT05255861
Title: An Exploratory Study of HRD Score in Chinese Ovarian Cancer Patients Benefiting From PARP Inhibitor Targeted Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xin Wu (Other)
Responsible Party: Sponsor-Investigator, Xin Wu, Department Director, Obstetrics & Gynecology Hospital of Fudan University
Organization: Obstetrics & Gynecology Hospital of Fudan University (Other)
Other Study IDs: FUOBGY2021-246
Record Dates: First submitted 2022-02-15; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
Keywords: Homologous Recombination Deficiency Score
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project intends to evaluate the sensitivity of different Homologous Recombination Deficiency (HRD) score to Poly(ADP-ribose) polymerase inhibitor (PARPi) by retrospectively analyzing the tissue samples of patients with ovarian cancer using PARPi, and to determine the cut off value of the HRD score algorithm suitable for the Chinese population, so as to provide evidence for the role of PARPi in ovarian cancer. The screening of the beneficiaries of maintenance therapy provides precise guidance and can be used as a reference for other cancer types.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. high-grade serous/endometrioid epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer;
3. FIGO stage III or IV;
4. at least 6 cycles and no more than 9 cycles First-line platinum-containing chemotherapy;
5. CR or PR after chemotherapy;
6. ECOG 0-1;
7. sufficient biological samples for HRD score detection;
8. patients signed informed consent;
9. good bone marrow function.

Exclusion Criteria:

1. incomplete follow-up records of survival information;
2. unqualified biological sample quality control

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese women with ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Homologous Recombination Deficiency score | After the ovarian tissue is obtained, an average of 3 year
  Optimize the Homologous Recombination Deficiency scoring algorithm to calculate the Homologous Recombination Deficiency score of each patient's ovarian cancer tissue

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wu, PHD, Principal Investigator — The Obstetrics and Gynecology Hospital of Fudan University
Locations (1):
- The Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No